CLINICAL TRIAL: NCT04049838
Title: Ultrasound Guided Posterior Versus Lateral Transversus Abdominis Plan Block for Prolonged Postoperative Analgesic Effect in Children . Randomized Controlled Trial
Brief Title: Ultrasound Guided Posterior Versus Lateral Transversus Abdominis Plan Block for Prolonged Postoperative Analgesic Effect in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Maher Kamel, lecture of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 011223456
Record Dates: First submitted 2019-07-21; First posted 2019-08-08 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lateral transversus abdominis block (Active Comparator): patients will take lateral transversus abdominis plan block. The block will be done unilaterally on the same side of proposed surery with 0.25% bupivacaine at a volume of 1 ml·kg-1
  Interventions: Procedure: postoperative analgesia for lower abdominal surgery in children
- posterior tansversus abodominis plane block (Active Comparator): patients will take posterior transversus abdominis plane block. The block will be done unilaterally on the same side of proposed surery with 0.25% bupivacaine at a volume of 1 ml·kg-1
  Interventions: Procedure: postoperative analgesia for lower abdominal surgery in children
- convential analgesia (Active Comparator): conventional analgesia in form of 1 micrograms. Kg-1 fentanyl and paracetamol 15 mg. Kg-1 suppositories
  Interventions: Procedure: postoperative analgesia for lower abdominal surgery in children

INTERVENTIONS:
Procedure: postoperative analgesia for lower abdominal surgery in children — compare lateral and posterior approaches of trannsversus abdominis plane block for analgesia after lower abdominal surgery in children

SUMMARY:
Ultrasound Guided Posterior Versus Lateral Transversus Abdominis Plan Block for Prolonged Postoperative Analgesic Effect in Children

DETAILED DESCRIPTION:
the investigators will compare the effect of posterior Transversus abdominis plan block versus the effect of lateral transversus abdominis plan bock regarding the duration of analgesia and patients satisfaction the study will be conducted on 69 children aged from 1 to 7 years presented for lower abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* children from 1- 7 years
* scheduled to undergo lower abdominal surgery

Exclusion Criteria:

* bleeding disorders
* emergency surgery
* skin lesion at site of needle insertion

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2019-02-16 (Actual); Primary Completion 2019-11-05 (Estimated); Study Completion 2019-12-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain assessment by the CHEOPS score | the first 24 hours postoperative
  Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) for Post-Op Pediatric Pain the score is based on 6 crtiteria:
  1. crying
  2. facial expression
  3. child verbal expression
  4. body positiion
  5. touching or grabbing at wound
  6. legs position criterion 1 is given a score of 1-3, criterion 2 and 3 are given score 0-2, criterion 4,5 and 6 are given a score 1-2 making the worst possible score 13 while the least possible score is 4.
  a total score of 6 or less indicates adequate analgesia

SECONDARY OUTCOMES:
heart rate | at 2,4,8,12 and 24 hours postoperative
  Measurement of heart rate (beats per minute)
Mean arterial blood pressure | at 2,4,8,12 and 24 hours postoperative
  Measurement of Mean arterial blood pressure ( mm Hg)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Aini, Cairo, Egypt